CLINICAL TRIAL: NCT01134874
Title: The Comparison of a Technology-Based System and an In-Person Behavioral Weight Loss Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John M. Jakicic, PhD (Other)
Responsible Party: Sponsor-Investigator, John M. Jakicic, PhD, Professor and Chair, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO09040121
Record Dates: First submitted 2010-05-25; First posted 2010-06-02 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard weight loss intervention (Experimental)
  Interventions: Behavioral: Standard weight loss intervention
- Standard weight loss intervention plus technology (Experimental)
  Interventions: Behavioral: Standard weight loss intervention plus technology
- Technology only (Experimental)
  Interventions: Behavioral: Technology only

INTERVENTIONS:
Behavioral: Standard weight loss intervention — In-person weight loss sessions, dietary intake prescription of 1200-1500 kcal per day, exercise progressing to 300 minutes per week.
  Arms: Standard weight loss intervention
Behavioral: Standard weight loss intervention plus technology — In-person weight loss sessions, dietary intake prescription of 1200-1500 kcal per day, exercise progressing to 300 minutes per week, plus technology to provide real-time feedback on energy expenditure, plus a website to log dietary intake.
  Arms: Standard weight loss intervention plus technology
Behavioral: Technology only — One intervention telephone call per month, dietary intake prescription of 1200-1500 kcal per day, exercise progressing to 300 minutes per week, plus technology to provide real-time feedback on energy expenditure, plus a website to log dietary intake.
  Arms: Technology only

SUMMARY:
The primary aim of this study is to compare the changes in body weight between a technology-based system, an in-person behavioral weight loss intervention, and a combination of both during a 12 month behavioral weight loss intervention in adults. Sedentary, healthy overweight and obese adults will be recruited to participate. Assessments will be conducted at 0, 6, and 12 months. This is a randomized trial in which participants will be randomized to one of three groups: standard behavioral weight loss (SBWL), standard behavioral weight loss plus technology (SBWL+TECH), and technology alone alone (TECH).

ELIGIBILITY:
Inclusion Criteria:

* ages of 21-55 years
* Body mass index (BMI) between 25-39.9 kg/m2

Exclusion Criteria:

* Currently pregnant, pregnant in the last 6 months, or plan on becoming pregnant in the next 6 months.
* Currently participating in regular exercise for over 60 minutes/week.
* Taking any medications that affect body weight or metabolism (e.g. synthroid).
* Have any physical limitations that would prevent exercise.
* Currently being treated for coronary heart disease, diabetes mellitus, hypertension, or cancer.
* Have a history of myocardial infarction or other heart-related surgeries.
* Have a resting systolic blood pressure > 150 mmHg or diastolic blood pressure of > 100 mmHg or currently taking any medications that affect blood pressure or heart rate (e.g. beta blockers).
* Currently enrolled in a commercial weight loss program, participating in another weight loss study, or in a weight loss study in the last 12 months.
* Have lost > 5% of current body weight in the past 6 months.
* Currently being treated for any psychological problems or taking any psychotropic medication.
* Currently do not have access to a computer and the Internet that can be used for this study. This requires a PC computer, the ability to load software for the technology system, an existing internet connection provided by the participant, and a dedicated USB port to allow the armband from the technology system to be connected to the computer for the download of information.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
weight | change from 0 to 6 months
  Body weight will be assessed on a digital scale to assess change in body weight over the intervention period.

SECONDARY OUTCOMES:
cardiorespiratory fitness | 0, 6, 12, months
  A graded exercise test on a treadmill along with indirect calorimetry will be used to measure cardiorespiratory fitness. This will provide a measure of oxygen consumption and metabolic equivalents of work at the time of test termination.
body composition | 0, 6, 12 months
  Body composition will be assessed using dual energy X-ray absorptiometry (DXA). This will provide a measure of lean body mass, fat mass, bone mineral content, and percent body fat.
physical activity | 0, 6, 12 months
  A questionnaire and a portable device worn on the upper arm will be used to measure and quantify energy expenditure from physical activity.
dietary intake | 0, 6, 12 months
  A questionnaire will be used to assess self-reported food intake. This will be used to estimate calories, dietary fat, protein, and carbohydrates consumed.
psychosocial and behavioral measures | 0, 6, 12 months
  Questionnaires will be used to assess self-efficacy for weight loss and physical activity, barriers to physical activity and weight loss, expected outcomes resulting from physical activity and weight loss, perceived body image, depressive symptomotology, weight history, dietary disinhibition and restraint, and behaviors typically related to weight loss (e.g., self-weighing, meal planning, etc.).
Weight change | weight at 0, 6, and 12 months
  Body weight measured on a digital scale

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Pittsburgh; Steve Verba, MS, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States